CLINICAL TRIAL: NCT06910397
Title: Evaluating The Effect of Probiotics on Oral Health Status and Its Influence on The Gingival Disease and Halitosis in Iraq
Brief Title: The Effect of Probiotics on Gums Health and Bad Breath
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Mustansiriyah University (Other)
Responsible Party: Principal Investigator, BAYDAA ABDULQAHAR YOUNUS, Principal Investigator, Al-Mustansiriyah University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MUPRV13
Record Dates: First submitted 2025-03-20; First posted 2025-04-04 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-02

CONDITIONS: Gingivitis
Keywords: probiotics and gingival health
MeSH Terms: conditions — Gingivitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- probiotic group (Active Comparator): each participant will take one tablet of probiotic daily for 28 days
  Interventions: Drug: Probiotic Arm
- placebo group- (Placebo Comparator): each participant will take one tablet of placebo tablet daily for 28 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Probiotic Arm — one tablet daily for 28 days
  Arms: probiotic group
Other: Placebo — placebo tablet once daily for 28 days
  Arms: placebo group-

SUMMARY:
the study is about using healthy bacteria to improve the overall gingival and overall health and prevent or decrease the bad odor of the mouth caused by bad bacteria

DETAILED DESCRIPTION:
The goal of this study is to verify the effect of Probiotics on oral Health Status and eliminate the gingival disease and Halitosis by measuring the levels of salivary biomarkers (cytokine IL-1b and proteases Matrix metalloproteinase (MMP-8) in saliva) and level of volatile sulfur compounds (VSCs) and their effects on improving gingival diseases clinical parameters in person age of (17-25) years old. The participants are randomly divided into two parallel groups (A, B). Group A will take probiotics and group B will take placebo for 28 days. The levels of IL-1b, MMP-8 in saliva, and VSCs measurement will be recorded respectively in different intervals of zero time and repeated on 14 days and 28 days.

Statistical analysis will be done then comparative between two groups

ELIGIBILITY:
The Inclusion criteria

* Subjects (male and female) between the age range 17-25 years old.
* Subjects with mouth breathing habit.
* Subjects with orthodontic and prosthodontic appliance
* Race from Iraq.
* Subjects having a dentition with ≥20 evaluable teeth (minimum of five teeth per quadrant).

The Exclusion criteria

* History of chronic disease.
* History of systemic disease.
* Patients with autoimmune diseases.
* Patients under antibiotic treatment.
* Pregnant, lactating females.
* History of undergoing nonsurgical and surgical periodontal therapy in the last 6 months.

Ages: 17 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 88 (Actual)
Dates: Start 2025-04-03 (Actual); Primary Completion 2025-05-03 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
oral health measures for 90 participant of both group | four weeks(0day,14 day,28 day)
  gingival index (scale 0-3),plaque index (scale 0-3), oral health index- simplex is composed of the Debris index and Calculus index (scoring six tooth segments in the mouth for each participants in both groups for the study and control group.
Halitosis (90 participant of both group) | four weeks(0 day,14 day, 28 day)
  Measuring the level of volatile sulfur compounds (VSCs) by use heliometer device (YRY Smart Breath Odor Detector), calculate social distance on (cm unite), detailed odor concentration on(ppm unite), and the related light color on the display screen for each participants in both groups the study and control group.

SECONDARY OUTCOMES:
The salivary biomarkers (90 participant of both group) | four weeks (0 day,14 day ,28 day)
  Pro-inflammatory cytokine IL-1B (pg/ml). Matrix metalloproteinase neutrophil collagenase MMP-8 (pg/ml) for each participants in both groups the study and control group.

CONTACTS AND LOCATIONS:
Overall Officials: BAYDAA Y Alani, MSc student, Principal Investigator
Locations (1):
- AL- Mustansiriyah University College of Dentistry, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-01-05): https://cdn.clinicaltrials.gov/large-docs/97/NCT06910397/ICF_000.pdf